CLINICAL TRIAL: NCT00359008
Title: PHP Preferential Hyperacuity Perimeter for the Detection of Choroidal Neovascularization (CNV)
Brief Title: PHP Home Preferential Hyperacuity Perimeter for the Detection of Choroidal Neovascularization (CNV)
Status: Completed | Type: Observational
Sponsor: Notal Vision Ltd. (Industry)
Responsible Party: Osnat Ehrman, NotalVision
Organization: Notal Vision Inc. (Industry)
Other Study IDs: PHP V3
Record Dates: First submitted 2006-07-30; First posted 2006-08-01 (Estimated); Last update posted 2008-01-15 (Estimated); Status verified 2008-01

CONDITIONS: Age Related Macular Degeneration
Keywords: AMD; CNV; PHP
MeSH Terms: conditions — Macular Degeneration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- 1: Intermediate AMD
- 2: New untreated CNV subject

SUMMARY:
The primary objective of this study is to assess the ability of the PHP & HPHP to detect newly diagnosed non treated Chorodial neovascularization (CNV) lesion associate with advanced age related Macular Degeneration (AMD) and differentiate them from Early/intermediate/GA AMD

DETAILED DESCRIPTION:
the study is prospective, multi-center, comparative

The PHP is a class I FDA approved Device ( K050350 )

ELIGIBILITY:
Inclusion Criteria:

* Patients with AMD related lesions:

Newly diagnosed (up to 6 months) non-treated CNV patients secondary to AMD in the study eye, or GA patients or Early and Intermediate AMD patients.

* Age ³ 50 for AMD patients
* VA with habitual correction in study eye 6/60 or better
* Mental and physical ability to perform a PHP/HPHP test
* Subject able and willing to sign consent form and participate in study
* Subject is not participating in another study when conducting the test

Exclusion Criteria:

* Evidence of macular disease other than AMD or Glaucoma in the study eye.

  * Presence of any significant media opacity that precludes a clear view of the macular area as identified by biomicroscopy, fundus photography, or fluorescein angiography in the study eye
  * Any non-macular related ocular surgery performed within 3 months prior to the study in the study eye
  * CNV patient inability to tolerate intravenous fluorescein angiography

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: At least 200 subjects with intermediate AMD in at least one (1) eye based on medical record review and/or clinical diagnosis and at least 200 subjects with neovascular AMD in at least one (1) eye in all sites.
Sampling Method: Probability Sample
Enrollment: 336 (Actual)
Dates: Start 2006-07; Study Completion 2007-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ofer Sharon, MD, Study Director — Notal Vision
Locations (1):
- Ha'emek Hospital, Afula, Israel

REFERENCES:
- [Background] Alster Y, Bressler NM, Bressler SB, Brimacombe JA, Crompton RM, Duh YJ, Gabel VP, Heier JS, Ip MS, Loewenstein A, Packo KH, Stur M, Toaff T; Preferential Hyperacuity Perimetry Research Group. Preferential Hyperacuity Perimeter (PreView PHP) for detecting choroidal neovascularization study. Ophthalmology. 2005 Oct;112(10):1758-65. doi: 10.1016/j.ophtha.2005.06.008. PMID 16154198
- [Background] Goldstein M, Loewenstein A, Barak A, Pollack A, Bukelman A, Katz H, Springer A, Schachat AP, Bressler NM, Bressler SB, Cooney MJ, Alster Y, Rafaeli O, Malach R; Preferential Hyperacuity Perimeter Research Group. Results of a multicenter clinical trial to evaluate the preferential hyperacuity perimeter for detection of age-related macular degeneration. Retina. 2005 Apr-May;25(3):296-303. doi: 10.1097/00006982-200504000-00008. PMID 15805906
- [Background] Bressler NM. Age-related macular degeneration is the leading cause of blindness.. JAMA. 2004 Apr 21;291(15):1900-1. doi: 10.1001/jama.291.15.1900. No abstract available. PMID 15108691
- [Background] Bressler NM. Early detection and treatment of neovascular age-related macular degeneration. J Am Board Fam Pract. 2002 Mar-Apr;15(2):142-52. PMID 12002198
- [Background] Enoch JM, Williams RA, Essock EA, Barricks M. Hyperacuity perimetry. Assessment of macular function through ocular opacities. Arch Ophthalmol. 1984 Aug;102(8):1164-8. doi: 10.1001/archopht.1984.01040030942019. PMID 6466179
- See also: Company Site — http://www.notalvision.com